CLINICAL TRIAL: NCT05149898
Title: Open-Label, Tolerability and Efficacy Study of ZYN002 Administered as a Transdermal Gel to Children and Adolescents With 22q11.2 Deletion Syndrome
Brief Title: Open-Label Study of ZYN002 Administered as a Transdermal Gel to Children and Adolescents With 22q11.2 Deletion Syndrome
Acronym: INSPIRE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zynerba Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYN2-CL-031
Record Dates: First submitted 2021-10-05; First posted 2021-12-08 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: 22Q Deletion Syndrome
Keywords: 22qDS; Chromosome 22q11.2 deletion syndrome; Autosomal dominant Opitz G/BBB syndrome; CATCH22; Cayler cardiofacial syndrome; Conotruncal anomaly face syndrome (CTAF); Shprintzen syndrome; Velo-cardio-facial syndrome (VCFS); Velocardiofacial syndrome
MeSH Terms: conditions — DiGeorge Syndrome; Cayler cardiofacial syndrome

STUDY DESIGN:
Intervention Model Description: Open-label study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label (Experimental): Open-label
  Interventions: Drug: ZYN002

INTERVENTIONS:
Drug: ZYN002 — CBD Transdermal Gel pharmaceutically manufactured. Cannabidiol (CBD) formulated as a clear gel (transdermal delivery).
  Dose received is based on weight.
  1. Patients who weigh ≤ 35 kg will receive 125 mg CBD Q12H (every 12 hours); for a total daily dose of 250 mg CBD.
  2. Patients who weigh > 35 kg will receive 250 mg CBD Q12H (±2 hours); for a total daily dose of 500 mg CBD.
  Other Names: Cannabidiol Transdermal Gel

SUMMARY:
To evaluate the safety and tolerability of ZYN002 administered as a transdermal gel formulation, for up to 38 weeks, in patients ages 4 to < 18 years, in the treatment of 22q.11.2 Deletion Syndrome (22qDS).

DETAILED DESCRIPTION:
This is an open-label study to assess the safety, tolerability and efficacy of cannabidiol (CBD) administered as ZYN002, a transdermal gel, for the treatment of child and adolescent patients with 22qDS. Male and female patients with 22qDS will be treated in Period 1 for 14 weeks. Patients that meet study criteria will be allowed to continue to Period 2 for an additional 24 weeks of treatment. At the end of study, patients taking antiepileptic drug (AED) medication(s) will have an additional one or two week Taper Period. Approximately 20 male and female patients, ages 4 to < 18 years, will receive ZYN002.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children and adolescents aged 4 to less than 18 years, at the time of Screening.
2. Judged by the Investigator to be in generally good health at Screening based upon the results of a medical history, physical examination, and clinical laboratory test results.
3. Patients must have a diagnosis of 22q Deletion Syndrome (22qDS) confirmed by genetic testing.
4. Patients have a Clinical Global Impression-Severity (CGI-S) score of 4 or higher at Screening and Visit 2.
5. Patients must have a Pediatric Anxiety Rating Scale-Revised (PARS-R) severity score of 10 or higher at Screening and Visit 2.
6. Patients with a history of seizure disorders must currently be receiving treatment with a stable regimen of one or two AEDs, or must be seizure-free for one year if not currently receiving AEDs.
7. If patients are receiving non-pharmacological behavioral and/or dietary interventions, they must be stable for three months prior to Screening.
8. Patient has demonstrated stable calcium levels for one year prior to Screening.
9. Patients have a body mass index between 12-35 kg / m2 (inclusive).
10. Females of childbearing potential must have a negative pregnancy test at the Screening Visit and a negative pregnancy test at all designated study visits.
11. Patients and parents/caregivers agree to abide by all study restrictions and comply with all study procedures.
12. Patients and parents/caregivers must be adequately informed of the nature and risks of the study and give written informed consent (and assent if applicable) prior to Screening.
13. Parents/caregiver(s) must provide written consent to assist in study drug administration.
14. In the Investigator's opinion, patients and parents/caregivers are reliable and willing and able to comply with all protocol requirements and procedures.

Exclusion Criteria:

1. Females who are pregnant, nursing, or planning a pregnancy; females of childbearing potential and male patients with a partner of childbearing potential who are unwilling or unable to use an acceptable method of contraception for the duration of therapy and for three months after the last dose of study medication.
2. History of significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to any compound or chemical class related to ZYN002 or its excipients.
3. Exposure to any investigational drug or device ≤ 30 days prior to Screening or at any time during the study.
4. Patient has ALT, AST, or total bilirubin levels ≥ 2 times the ULN)or has alkaline phosphatase levels ≥ 3 times the ULN as determined from Screening safety laboratories.
5. Use of cannabis or any THC or CBD-containing product within three months of Screening Visit or during the study.
6. Patient has a positive drug screen.
7. Patient is using the following AEDs: clobazam, phenobarbital, ethosuximide, felbamate, carbamazepine, phenytoin or vigabatrin.
8. Patient is using any strong inhibitor/inducer of CYP3A4 or sensitive substrate for CYP3A4 including but not limited to the following medications: midazolam, oral ketoconazole, fluconazole, nefazadone, rifampin, alfentanil, alfuzosin, amiodarone, cyclosporine, dasatinib, docetaxol, eplerenone, ergotamine, everolimus, fentanyl, halofantrine, irinotecan, lapatinib, levomethadyl, lumefantrine, nilotinib, pimozide, quinidine, ranolazine, sirolimus, tacrolimus, temsirolimus, toremifene, tretinioin, vincristine, vinorelbine, St. John's Wort, and grapefruit juice/products.
9. Patient with diagnosis of known genetic disorder, other than 22qDS.
10. Patient has diagnosis of DiGeorge or Velocardiofacial syndrome without the presence of 22qDS.
11. Patient has a primary psychiatric diagnosis other than 22qDS or anxiety, including bipolar disorder, psychosis, schizophrenia, PTSD or major depressive disorder.
12. Patient is on stable treatment of >6 months of not more than two psychoactive medications at screening or throughout the study (with the exception of one psychoactive medication prescribed for sleep).
13. Patient has an advanced, severe, or unstable disease that may interfere with the study outcome evaluations.
14. Patient is expected to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
15. Patient has an acute or progressive neurological disease, or any psychiatric disorder or severe mental abnormalities that are likely to require changes in drug therapy or interfere with the objectives of the study or ability to adhere to protocol requirements.
16. Patient has a positive result for the presence of HBsAg, HCV, or HIV antibodies.
17. Patients at risk of needing cardiovascular surgical repair within the upcoming 12 months.
18. Patient has unstable cardiovascular disease, such as advanced arteriosclerosis, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, cardiac conduction problems, exercise-related cardiac events including syncope and pre-syncope, risk factors for Torsades de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome), other serious or other clinically unstable cardiac problems as indicated by history, physical examination, or ECG.
19. Any clinically significant condition or abnormal findings at the Screening Visit that would, in the opinion of the Investigator, preclude study participation or interfere with the evaluation of the study medication.
20. Any skin disease or condition that may affect treatment application, application site assessments, or absorption of the study drug.
21. History of treatment for, or evidence of, drug abuse within the past year.
22. Patient responds "yes" to Question '4' or '5' on the Columbia Suicide Severity Rating Scale Children (C-SSRS) during Screening or at any time on study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | Adverse Event time frame is from admission to a study completion, an average of 9 months
  Safety assessment will include collection of any treatment-emergent adverse events (safety and tolerability).

SECONDARY OUTCOMES:
Aberrant Behavior Checklist (ABC-C) Pre-specified Subscale 1 | Screening, Visit 2, Visit 3, Visit 4, Visit 5, Visit 6, and Visit 7 EOS/ET, over a 38 week period
  ABC-C is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials.
Clinical Global Impression-Severity and Improvement (CGI-S and CGI-I) | CGI-S is collected at Screening, Visit 2, Visit 3, Visit 4, Visit 5, Visit 6, and Visit 7 EOS/ET, over a 38 week period and CGI-I will be assessed at Visit 3 and Visit 4/EOS/ET, over 14 week period
  CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  CGI-I is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a Baseline state at the beginning of the intervention and rated as: 1 - very much improved; 2 - much improved; 3 - minimally improved; 4 - no change; 5 - minimally worse; 6 - much worse; or 7 - very much worse.
Anxiety, Depression and Mood Scale (ADAMS) | Screening, Visit 2, Visit 3, Visit 4, Visit 5, Visit 6, and Visit 7 EOS/ET, over a 38 week period
  The ADAMS is comprised of 28 items, which are rated on a scale of "0 - not a problem" to "3 - severe problem." The ADAMS yields a total score as well as five subscale scores: "Manic/Hyperactive Behavior," "Depressed Mood," "Social Avoidance," "General Anxiety," and "Compulsive Behavior."
Qualitative Caregiver Reported Behavioral Problems Survey | Visit 3, Visit 4, Visit 5, Visit 6, and Visit 7 EOS/ET, over a 38 week period
  The parent/caregiver will be asked the following question "What are the three behavioral, emotional, or social problems that most impacted your son/daughter and his/her family in approximately the past year?" At each study visit the parent/caregiver will be reminded of their responses from the Screening Visit in order to rate the three questions for improvement or worsening.
Pediatric Anxiety Rating Scale-Revised (PARS-R) | Screening, Weeks 14, 22, 30, and Week 38
  The PARS-R is a clinician-rated caregiver interview that covers 61 behaviors related to anxiety. The PARS-R provides broad coverage of separation anxiety, social phobia, and generalized anxiety. Symptoms are further categorized into Social Interactions or Performance Situations, Separation, Generalized, Specific Phobia, Panic Symptoms/Physical Signs, Obsessive-Compulsive, Health/Illness Concerns, and Other.

CONTACTS AND LOCATIONS:
Overall Officials: Carol O'Neill, Study Director — VP, Development
Locations (3):
- Greenwood Genetic Center, Greenville, South Carolina, United States
- Australia (2):
  - Lady Cilento Children's Hospital - South Brisbane, Brisbane, Queensland
  - Genetics Clinics Australia, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.